CLINICAL TRIAL: NCT05272683
Title: An Open-label, Fixed-sequence, Drug-drug Interaction Study in Healthy Subjects to Evaluate the Effect of Itraconazole, a Strong CYP3A4 Inhibitor and Potent P-gp Inhibitor on the Pharmacokinetics of GLPG3667
Brief Title: Drug-drug Interaction Study with GLPG3667 and Itraconazole in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GLPG3667-CL-109
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-05

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GLPG3667 + itraconazole (Experimental)
  Interventions: Drug: GLPG3667; Drug: Itraconazole

INTERVENTIONS:
Drug: GLPG3667 — On day 1 and day 8, participants will receive a single dose
Drug: Itraconazole — On days 5 to 11, participants will receive itraconazole once daily

SUMMARY:
The main purpose of this study is to determine the effect of itraconazole on the amount of GLPG3667 that gets into the blood when the 2 drugs are administered together compared to when GLPG3667 is administered alone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 55 years of age (extremes included), on the date of signing the informed consent form (ICF). Female subjects should be of non-childbearing potential, defined as permanently surgically sterile (bilateral oophorectomy, i.e. surgical removal of ovaries, bilateral salpingectomy or hysterectomy, i.e. surgical removal of uterus), or with no menses for 12 or more months without an alternative medical cause AND a follicle-stimulating hormone (FSH) level in the postmenopausal range. For surgical sterilization, documented confirmation will be requested.
* A body mass index between 18.0 and 30.0 kg/m2, inclusive.
* Judged to be in good health by the investigator based upon the results of a medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and fasting clinical laboratory safety tests. Neutrophil, lymphocyte, and platelet counts must be above the lower limit of normal range. Total bilirubin, aspartate aminotransferase (AST), and alanine aminotransferase (ALT) must be within normal ranges. Other clinical laboratory safety test results must be within the normal ranges or test results that are outside the normal ranges need to be considered not clinically significant in the opinion of the investigator.

This list only contains the key inclusion criteria.

Exclusion Criteria:

* Known hypersensitivity to ingredients of GLPG3667 and/or itraconazole, or history of a significant allergic reaction to ingredients of GLPG3667 and/or itraconazole, as determined by the investigator.
* Treatment with any medication (including over-the-counter (OTC) and/or prescription medication, dietary supplements, nutraceuticals, vitamins and/or herbal supplements, and hormonal replacement therapy) except occasional paracetamol (maximum dose of 2 g/day and maximum of 10 g/2 weeks) in the last 2 weeks or 5 half-lives of the drug, whichever is longer, prior to the first dosing.

This list only contains the key exclusion criteria.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of GLPG3667 | From Day 1 pre-dose until Day 12
  To determine the effect of itraconazole on the pharmacokinetics (PK) of GLPG3667
Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) of GLPG3667 | From Day 1 pre-dose until Day 12
  To determine the effect of itraconazole on the PK of GLPG3667

SECONDARY OUTCOMES:
Frequency and severity of treatment-emergent adverse events (TEAEs), treatment-emergent serious adverse events (SAEs), and TEAEs leading to treatment discontinuation. | From Day 1 through study completion, an average of 2 months
  To evaluate the safety and tolerability of GLPG3667 alone or when co-administered with itraconazole

CONTACTS AND LOCATIONS:
Overall Officials: Galapagos Study Director, MD, Study Director — Galapagos NV
Locations (1):
- Altasciences, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No